CLINICAL TRIAL: NCT05401461
Title: Does Mobilisation in the Evening Reduce the Incidence of Delirium in Patients Admitted to Intensive Care: a Mixed-methods, Randomised Controlled Feasibility Study
Brief Title: Mobilisation in the EveNing to TreAt Delirium
Acronym: MENTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW584022
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Critical Illness; Sleep Disturbance; Mobility Limitation; Intensive Care Unit Delirium
Keywords: delirium; non-pharmacological; mobilisation; sleep; intensive care; ICU
MeSH Terms: conditions — Critical Illness; Parasomnias; Mobility Limitation; Delirium

STUDY DESIGN:
Intervention Model Description: Mixed methods, randomised controlled feasibility study
Who Masked: Investigator, Outcomes Assessor
Masking Description: All outcomes will be collected by an independent researcher blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Evening mobilisation delivered between 7pm and 9pm
  Interventions: Other: Evening mobilisation
- Control (No Intervention): Patients in the control arm will receive standard care which incorporates physiotherapy and mobilisation as appropriate between 8am and 5pm

INTERVENTIONS:
Other: Evening mobilisation — Evening mobilisation delivered between (19.00 and 21.00) according to standardised procedures and established safety criteria. The intervention will begin on day 1 of admission or the first evening following recruitment. Mobilisation will be defined as a score of ≥ 2 on the Manchester mobility score (sit on the edge of the bed or higher), with actual mobilisation level achieved and duration of intervention based on clinical decision of the mobilisation therapists. Patients will also be offered the opportunity to engage in activities which may be part of their normal evening routines (e.g. brushing teeth, reading or watching television). The intervention will be carried out for up to seven consecutive evenings. The evening mobilisation will be delivered in addition to any input from the MDT during normal daily working hours and will not replace any standard therapy.
  Arms: Intervention

SUMMARY:
Patients with severe illness require lifesaving treatment in intensive care units. Around a third of patients admitted to intensive care develop delirium. This is a severe state of confusion. Delirium can be a frightening experience. Patients suffering from delirium can find it difficult to think clearly or understand what is happening. In some cases delirium can cause people to see or hear things that are not really there. Patients who develop delirium tend to spend longer in hospital and have worse overall outcomes. A major cause for the development of delirium is poor sleep. Previous research suggests that delirium levels can be reduced when patients are more active. The investigators have noticed that when patients in intensive care have physiotherapy during the day, they are often very tired and fall asleep quickly afterwards. The investigators think that patients who have physiotherapy in the evening will sleep better overnight and hope this will subsequently reduce the number who develop delirium.

To answer this question the investigators need to compare patients who are active in the evening with those who only have physiotherapy sessions during the day. Before a full study can take place it is important to make sure it is designed in the best way. To do this, 60 patients will be recruited from 2 hospitals in the UK over 6 months. Half of those who agree to take part will be seen by the physiotherapist in the evening, the other half will not. The investigators will then ask the following questions before deciding whether to do a full study

1. Will patients agree to be a part of this trial?
2. Will they agree to the additional physiotherapy sessions offered in the evening?
3. Will patients and staff members be happy for us to randomly select who receives this extra treatment?

DETAILED DESCRIPTION:
The investigators hypothesise that mobilisation in the evening will promote more natural sleep, with patients becoming tired from physical exertion and plan to evaluate the impact this may have on reducing the incidence or duration of delirium.

A mixed-methods, two centre, randomised controlled feasibility study to establish the viability of conducting a larger multicentre RCT to test the effects of evening mobilisation on the incidence of ICU-acquired delirium.

Part 1 will evaluate whether it is possible to achieve acceptable recruitment and retention rates, intervention fidelity, and if the proposed data collection methods are appropriate.

Part 2 includes an acceptability analysis and qualitative evaluation, aiming to explore both patient and staff subjective experiences of the study intervention and proposed research methods (including willingness for randomisation and study outcome measures) and provide information to refine the study intervention (if required). The investigators will use principles of Normalisation Process Theory [28] and the NoMAD assessment tool [29] to assess the practicalities associated with implementing additional evening physiotherapy.

Treatment / Intervention The intervention will be delivered by a dedicated mobilisation team recruited from the study centres and will include trained ICU physiotherapists. Mobilisation will be delivered according to standardised procedures and established safety criteria. The intervention will begin on day 1 of admission or the first evening following recruitment.

After consultation with the responsible physician and nurse, patients will be approached between 19.00 and 21:00 to confirm suitability and consent to mobilise. Patients who are asleep will not be woken for the intervention. Mobilisation will be defined as a score of ≥ 2 on the Manchester mobility score (sit on the edge of the bed or higher), with actual mobilisation level achieved and duration of intervention based on clinical decision of the mobilisation therapists. Patients will also be offered the opportunity to engage in activities which may be part of their normal evening routines (e.g. brushing teeth, reading or watching television).

The intervention will be carried out for up to seven consecutive evenings. The intervention will be terminated if a) patient condition deteriorates irretrievably and physiotherapy is no longer appropriate, b) after seven evenings, or c) when the patient is discharged from the ICU. The intervention will not continue at secondary wards or units.

The evening mobilisation will be delivered in addition to any input from the MDT during normal daily working hours and will not replace any standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Admitted to ICU,
* Able to respond to verbal stimulus (Richmond Agitation Sedation Scale ≥ -3)
* Expected to stay in the ICU for at least 24 hours.

Exclusion Criteria:

* Death expected within the next 72 hours,
* Immobility prior to admission,
* Mobilisation contraindicated (e.g., spinal injury),
* Delirium diagnosis during this ICU admission,
* Acute or subacute severe neurological deficit or injury;
* Severe psychiatric illness (not including depression) or developmental problems;
* Suspected or confirmed drug or alcohol intoxication/overdose or withdrawal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 3 month recruitment window
  Proportion of patients agreeing to take part out of all those invited
Retention rate | Up to 7 days following recruitment
  Proportion of participants who complete the intervention
Intervention fidelity | Up to 7 days following recruitment
  Percentage of intervention sessions completed

SECONDARY OUTCOMES:
Incidence of delirium | During critical care stay, average of 2 weeks
  Incidence of delirium assessed as a positive result on the CAM-ICU
Duration of delirium | During critical care stay, average of 2 weeks
  counted at 12-hour periods; the end of delirium is defined when patients are delirium-negative for 24h or discharged to the ward
Sleep quality | During critical care stay, average of 2 weeks
  as an average and assessed over time using the Richard Campbell Sleep Questionnaire. This provides a score from 0 - 60, with higher scores representing better quality of sleep
Mobility level at critical care discharge | At ICU discharge, average of 2 weeks
  Assessed using the Manchester mobility score. Scores range from 1-7 with higher scores representing higher levels of mobility

CONTACTS AND LOCATIONS:
Overall Officials: David McWilliams, PhD, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (2):
- United Kingdom (2):
  - University Hospitals Coventry & Warwickshire, Coventry, Midlands
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McWilliams DJ, King EB, Nydahl P, Darbyshire JL, Gallie L, Barghouthy D, Bassford C, Gustafson OD. Mobilisation in the EveNing to prevent and TreAt deLirium (MENTAL): a mixed-methods, randomised controlled feasibility trial. EClinicalMedicine. 2023 Jul 19;62:102101. doi: 10.1016/j.eclinm.2023.102101. eCollection 2023 Aug. PMID 37533416
- [Derived] McWilliams D, King E, Nydahl P, Darbyshire JL, Gallie L, Barghouthy D, Bassford C, Gustafson O. Mobilisation in the EveNing to TreAt deLirium (MENTAL): protocol for a mixed-methods feasibility randomised controlled trial. BMJ Open. 2023 Feb 3;13(2):e066143. doi: 10.1136/bmjopen-2022-066143. PMID 36737097